CLINICAL TRIAL: NCT05185570
Title: Evaluation of the Risk Factors Influencing the Prognosis of Elderly Patients With Acute Poisoning.
Brief Title: Prognosis of Elderly Patients With Acute Poisoning.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Abeer hussien Mohamed, Teaching assistant in Forensic Medicine &Clinical Toxicology Department Faculty of Medicine, Sohag University
Other Study IDs: Soh-Med-21-12-01
Record Dates: First submitted 2021-12-12; First posted 2022-01-11 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2021-12

CONDITIONS: Acute Poisoning

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Acute poisoning is a major public health problem all over the world, it causes significant mortality and morbidity. It primarily involves younger populations, with less than 3% of the affected cases being in people aged 60 years or older in most studies. More than half of the intoxication events in the elderly over 65 years old were accidental.

DETAILED DESCRIPTION:
The elderly are different from younger adults in many aspects. There are age related physiological changes. They have a higher incidence of comorbidities and use of many medications for chronic conditions, both of which make the elderly more susceptible to acute poisoning and its related consequences.

Although the elderly form a relatively small proportion of those admitted to hospital for acute self-poisoning, the poisoning in them is often more serious, complications are more frequent and a fatal outcome is more common.

The presence of multiple physical, social, and psychiatric problems, with possible difficulties in the diagnosis of poisoning make the management of the elderly more complicated than that of younger poisoned patients. There are three main difficulties in diagnosing acute poisoning in the elderly. At first, it may not be easily obvious that the patient has taken an overdose. Secondly, the presence of pre-existing diseases may obscure the clinical picture and finally, the drug may cause physical signs that similar to common problems of old age.

ELIGIBILITY:
Inclusion Criteria:

all patients more than 60 years will be included.

Exclusion Criteria:

younger than 60 years.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: elderly patients with acute poisoning.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-01 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Change in Acute physiology and chronic health evaluation II score (APACHE II) in cases of elderly patients with acute poisoning. | 24 hours after admission to intensive care unit (ICU).
  "Acute Physiology And Chronic Health Evaluation II(APACHE II) " is a severity-of-disease classification system. one of several ICU scoring systems. It is applied within 24 hours of admission of a patient to an intensive care unit (ICU): an integer score from 0 to 71 is computed based on several measurements; higher scores correspond to more severe disease and a higher risk of death.
Change in Poisoning Severity Score (PSS) in cases of elderly patients with acute poisoning. | 24 hours after admission to intensive care unit (ICU).
  "Poisoning Severity Score (PSS)" is a standardized scale for grading the severity of poisoning allows qualitative evaluation of. morbidity caused by poisoning, better identification of real risks and comparability of data.